CLINICAL TRIAL: NCT02838173
Title: Serratus Plane Block for the Prevention of Chronic Pain After Breast Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Céline Boudart, MD, Erasme University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B406201628750
Record Dates: First submitted 2016-06-30; First posted 2016-07-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-06

CONDITIONS: Breast/Surgery; Postoperative Complication; Chronic Pain
MeSH Terms: conditions — Postoperative Complications; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- SPB (Experimental): Serratus Plane Bloc with Ropivacaine 2mg/ml (0,3ml/kg) and tissue infiltration with placebo made once, by the anesthetist in the operating theater before surgical incision
  Interventions: Procedure: serratus plane bloc : Ropivacaine 2mg/ml (0,3ml/kg); Procedure: tissue infiltration : placebo
- tissue infiltration (Active Comparator): tissue infiltration with Ropivacaine 2mg/ml (0,3ml/kg) and Serratus Plane Bloc with placebo made once, by the anesthetist in the operating theater before surgical incision
  Interventions: Procedure: tissue infiltration : Ropivacaine 2mg/ml (0,3ml/kg); Procedure: serratus plane bloc : placebo

INTERVENTIONS:
Procedure: serratus plane bloc : Ropivacaine 2mg/ml (0,3ml/kg)
  Arms: SPB
Procedure: tissue infiltration : Ropivacaine 2mg/ml (0,3ml/kg)
  Arms: tissue infiltration
Procedure: serratus plane bloc : placebo
  Arms: tissue infiltration
Procedure: tissue infiltration : placebo
  Arms: SPB

SUMMARY:
This study compare the "Serratus block plane" (SPB) and the local infiltration of the tissue in the prevention of acute and chronic pain after breast cancer surgery.

DETAILED DESCRIPTION:
Chronic pain after breast surgery may be severe, often requiring the use of morphine. The incidence of chronic pain varies from 27 to 50% depending on definitions.

The infiltration of tissues by a local anesthetic is a simple, fast and low risk technique but of limited effectiveness.

Serratus the flat block, performed under ultrasound guidance, is minimally invasive and easy to perform. It allows anesthesia and analgesia to an extended part of the anterolateral chest wall and the axilla. This regional anesthesia technique provides good analgesia during and after breast surgery, but remains to be evaluated; beyond perioperative analgesia, the benefit-risk, post operative rehabilitation, and the impact on ambulatory and on chronic pain are fundamental objectives.

ELIGIBILITY:
Inclusion Criteria:

* Women scheduled for elective breast neoplasm surgery
* Of ASA classification 1, 2 or 3
* Patients who provide written informed consent

Exclusion Criteria:

* Minor patients
* Patients refusing to sign the consent
* Patients included in another protocol within 3 months
* Pregnant or lactating patients
* Patients with history of allergy to local anesthetics (Ropivacaine)
* Patients with contraindication to regional anesthesia (coagulopathy, local infection ...)
* Patients with history of prior breast surgery (excluding diagnostic biopsy)
* Patients with history of chronic pain
* Patients with a history of psychiatric disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
postoperative chronic pain assessed using the DN4 questionnaire | 3 months postoperative
  DN4 questionnaire

SECONDARY OUTCOMES:
postoperative acute pain | day 1, day 2, day 3 postoperative
  Visual analogue scale (V.A.S.)
morphine consumption | day 1, day 2, day 3 postoperative

OTHER OUTCOMES:
length of stay in the Postoperative Acute Care Unit | through study completion
length of stay in hospital | through study completion

CONTACTS AND LOCATIONS:
Overall Officials: Luc Van Obbergh, MD PhD, Study Director — Erasme University Hospital

REFERENCES:
- [Background] Blanco R, Parras T, McDonnell JG, Prats-Galino A. Serratus plane block: a novel ultrasound-guided thoracic wall nerve block. Anaesthesia. 2013 Nov;68(11):1107-13. doi: 10.1111/anae.12344. Epub 2013 Aug 7. PMID 23923989
- [Background] Andreae MH, Andreae DA. Regional anaesthesia to prevent chronic pain after surgery: a Cochrane systematic review and meta-analysis. Br J Anaesth. 2013 Nov;111(5):711-20. doi: 10.1093/bja/aet213. Epub 2013 Jun 28. PMID 23811426